CLINICAL TRIAL: NCT05628181
Title: A Patient-facing Tool to Reduce Opioid-Psychotropic Polypharmacy in People Living With Dementia
Brief Title: A Patient-facing Tool to Reduce Opioid-Psychotropic Polypharmacy in People Living With Dementia (PLWD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Donovan Maust, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00218048; 3U54AG063546-03 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Polypharmacy; Dementia
Keywords: Central Nervous System medication; Education
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: There will be a total of four primary care clinics at University of Michigan Health and Henry Ford Health; potentially more clinics will be engaged if necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No educational tool (No Intervention): This arm will collect data on total standardized daily dosage of the medication classes contributing to CNS polyRx from the Electronic Medical Record (EMR).
- Educational nudge intervention (Experimental): Participants will be mailed the educational tool in the form of a brochure.
  Interventions: Behavioral: Educational nudge intervention

INTERVENTIONS:
Behavioral: Educational nudge intervention — This project will adapt the EMPOWER educational brochure for PLWD receiving CNS polyRx. The educational brochure will be mailed to intervention participants identified through EHR at Michigan Medicine and Henry Ford Health System. The brochure will describe what CNS polyRx is, present information about the associated risks, and suggest that participants speak with the prescribing clinician or pharmacist about ways to potentially simplify the medication regimen. The tool will be adapted through three successive rounds of focus groups (AIM one of this project) of PLWD.
  Arms: Educational nudge intervention

SUMMARY:
The goal of this project is to address central nervous system-active polypharmacy (CNS polyRx) in people living with dementia (PLWD) through focus groups and an educational intervention.

The project included three interconnected aims and engaged PLWD, care partners (CP), and clinicians. Aim 1 consisted of focus group discussions with PLWD and CPs, conducted to inform the development of the educational intervention. This aim was not considered a clinical trial. Therefore, this registration covers Aims 2 and 3, which constitute the clinical trial components. These included mailing the educational "nudge" intervention to PLWD and conducting qualitative interviews with clinicians. No care partners were involved in Aims 2 and 3.

The study hypothesizes that the total standardized daily dosage (TSDD) of medication classes contributing to CNS polyRx will decrease from baseline to 4 months among participants receiving the intervention.

DETAILED DESCRIPTION:
The United States (U.S.) health care system is poorly equipped to deal with the growing number of persons living with dementia (PLWD) in the U.S. and their complex medical and psychosocial needs. While memory impairment is the cardinal feature of Alzheimer's disease and related dementias (ADRD), behavioral and psychological symptoms (e.g., apathy, delusions, agitation) are common during all stages of illness and cause significant caregiver distress. CNS polyRx, defined by the American Geriatrics Society Beers Criteria as overlapping use of greater than or equal to (≥) 3 medications from any of the following six classes: antidepressants, antipsychotics, anti-epileptics, benzodiazepines, non-benzodiazepine benzodiazepine receptor agonist hypnotics, or opioids. CNS polyRx is common among PLWD with limited evidence to support such prescribing despite significant evidence of harms-an example of routine care provided to PLWD that is potentially harmful in the vast majority of cases.

Minimizing CNS polypharmacy is a critical opportunity to improve safe medication use for PLWD. Direct-to-patient education has been demonstrated as one successful approach to initiate deprescribing in older adults. For this pilot study, after developing the tool (Aim 1), the study team used the electronic health records (EHR) of two healthcare systems (UM and Henry Ford) to identify PLWD with CNS polypharmacy and sent the educational tool to these individuals. EHR review was then conducted to determine the implementation outcome of whether the recipients' clinicians were engaged in a discussion about these specific prescriptions. Finally, in preparation for a pragmatic trial, the study team queried the EHR to assess change in CNS-active prescribing in the months following receipt of the tool. The data generated during this pilot will allow the study team to seek future funding for a pragmatic trial to test this nudge intervention to reduce CNS polypharmacy among PLWD.

Note: While this project included three aims, only Aims 2 and 3 involved intervention activities and are included in this record. Aim 1, which involved qualitative focus groups with PLWD and their CP to inform the intervention's development, was exploratory in nature, did not constitute an intervention, and is therefore not included in this record. No care partners were involved in Aims 2 and 3 and are not included in this record.

This pragmatic trial of a clinic-level intervention received a waiver of informed consent. There is no informed consent document for the intervention. Clinicians from intervention clinics were interviewed to explore their perceptions about the acceptability of the experimental intervention only. No clinicians received an intervention, and no primary or secondary outcomes were planned based on these interviews.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are receiving care at the one of the selected primary care clinics at Michigan Medicine and Henry Ford Health System
* Individuals who have a diagnosis of dementia or mild cognitive impairment (MCI) of any type based on International Classification of Diseases (ICD-10) codes
* Individuals who have been prescribed ≥3 of the medications that contribute to CNS polyRx (e.g., antidepressants, antipsychotics, anti-epileptics, benzodiazepines, non-benzodiazepine benzodiazepine receptor agonist hypnotics, or opioids) based on chart review

Exclusion Criteria:

- primary care clinicians review of participants and determines intervention is not appropriate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donovan Maust, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett NM, Vordenberg SE, Kim HM, Turnwald M, Strominger J, Leggett AN, Akinyemi E, Blow FC, Vanderziel A, Pappas C, Maust DT. An Educational Intervention to Promote Central Nervous System-Active Deprescribing in Dementia: A Pilot Study. Drugs Aging. 2025 Mar;42(3):257-265. doi: 10.1007/s40266-024-01178-x. Epub 2025 Jan 20. PMID 39832105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinicians from intervention clinics were interviewed to assess their perceptions about the acceptability of the experimental intervention.
Pre-assignment Details: Individuals in the Clinicians arm did not receive an intervention.
Groups:
- No Educational Tool: Participants (PLWD) who did not receive the mailed the educational tool in the form of a brochure.
  This arm will collect data on total standardized daily dosage of the medication classes contributing to CNS polyRx from the Electronic Medical Record (EMR).
- Educational Nudge Intervention: Participants (PLWD) will be mailed the educational tool in the form of a brochure.
  Educational nudge intervention: This project will adapt the EMPOWER educational brochure for PLWD receiving CNS polyRx. The educational brochure will be mailed to intervention participants identified through EHR at Michigan Medicine and Henry Ford Health System. The brochure will describe what CNS polyRx is, present information about the associated risks, and suggest that participants speak with the prescribing clinician or pharmacist about ways to potentially simplify the medication regimen. The tool will be adapted through three successive rounds of focus groups (AIM one of this project).
- Clinicians: Clinicians from intervention clinics were interviewed to assess their perceptions about the acceptability of the experimental intervention.
Period: Overall Study
Arm/Group | No Educational Tool | Educational Nudge Intervention | Clinicians
Started | 68 | 61 | 10
Completed | 66 | 57 | 10
Not Completed | 2 | 4 | 0
Not completed — Death | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinicians: Clinicians who were interviewed but were not randomized to an intervention.
- Total: Total of all reporting groups
Arm/Group | No Educational Tool | Educational Nudge Intervention | Clinicians | Total
Number analyzed (Participants) | 61 | 68 | 10 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.4) | 73.7 (10.7) | 45.2 (10.7) | 63.3 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 8 | 89
  Male | 21 | 27 | 2 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 4 | 11 | 0 | 15
  White | 56 | 53 | 6 | 115
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 68 | 10 | 139

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Standardized Daily Dosage (TSDD) of CNS-Active Medications From Baseline to 4 Months, as Measured in the EHR
Description: CNS-polyRx included multiple meds from different classes. To track prescribing changes total standardized daily dosage (TSDD) unit is used. TSDD was calculated by dividing each med's prescribed daily dose by its Minimal Effective Geriatric Daily Dose (MEGDD) a framework for identifying the lowest effective daily dose for older adults to balance benefit and reduce harm. E.g., citalopram 20mg daily with MEGDD of 10mg=2 TSDD units. TSDD was assessed during 2 periods: 45day baseline and 45days before the 4month follow-up. For each period, the total supply of each CNS-active med was summed and divided by 45 days to get a daily dose, then divided by MEGDD to yield standardized daily dose for each med. Values were summed to get total TSDD/ participant. Primary outcome is change in TSDD, calculated as TSDD at 4months minus baseline TSDD. E.g.,45day supply of citalopram 20mg daily (MEGDD=10mg)=2, gabapentin 300mg TID (MEGDD=900mg)=1, and zolpidem 5mg daily (MEGDD=5mg)=1, results in TSDD of 4.0
Time Frame: Baseline (i.e., the 45 days prior to intervention) and 4 months post-intervention (i.e., the final 45 days of the 4-month period)
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | No Educational Tool | Educational Nudge Intervention
Number analyzed (Participants) | 68 | 61
doses per day
  TSDD At Baseline | 9.0 (7.2) | 9.0 (7.2)
  TSDD at 4 months | -1.3 (5.8) | -1.6 (6.0)

ADVERSE EVENTS:
Time Frame: 4 Months
Description: The intervention period was 4 months (i.e., potential prescription medication changes were examined 4 months after sending the educational intervention), during which time adverse events, including deaths, were also assessed. A final retrospective analysis at study completion (Aug 2024) captured any deaths during the intervention period that were not available in the EHR at the time of initial review. No adverse event data were collected from clinicians, as they did not receive an intervention.
Arm/Group | No Educational Tool | Educational Nudge Intervention | Clinicians
All-Cause Mortality (participants affected / at risk) | 2/68 | 4/61 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/68 | 4/61 | 0/0
Other Adverse Events (participants affected / at risk) | 0/68 | 0/61 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Educational Tool (N=68) | Educational Nudge Intervention (N=61) | Clinicians (N=0)
Death (General disorders) | 2 (2) | 4 (4) | 0 — Death/hospitalization can reasonably be expected considering the study population includes PLWD and those experiencing CNS polyRx, however, the study team does not have access to details related to the participant's cause of death.

LIMITATIONS AND CAVEATS:
The primary limitation of this pilot study was that it was conducted with a small number of PLWD at two health systems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT05628181/Prot_SAP_000.pdf